CLINICAL TRIAL: NCT05954897
Title: Lenvatinib, Tislelizumab Combined With RALOX Regimen HAIC in Advanced Hepatocellular Carcinoma: a Phase II, Single-arm, Prospective Study
Brief Title: Lenvatinib, Tislelizumab Combined With RALOX Regimen HAIC in Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-124-02
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Lenvatinib, Tislelizumab Combined with RALOX Regimen HAIC

INTERVENTIONS:
Drug: Lenvatinib, Tislelizumab Combined with RALOX Regimen HAIC — RALOX Regimen of Hepatic Arterial Infusion Chemotherapy (HAIC) Combine Lenvatinib and Tislelizumab

SUMMARY:
To evaluate the efficacy and safety of lenvatinib, tislelizumab combined with RALOX regimen HAIC in advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. HCC was diagnosed according to the Criteria for Diagnosis and Treatment of Primary Liver Cancer (2022 Edition) and American Association for the Study of Liver Diseases (AASLD) criteria.
3. Classified as stage C according to the Barcelona Clinic Liver Cancer (BCLC) staging system.
4. A dominant mass in theliver with or without extrahepatic oligometastasis, which was defined as up to three metastatic lesions in up to two organs with the largest diameter of≤3 cm.
5. No prior treatment for HCC.
6. At least one measurable target lesion according to modified Response Evaluation Criteria in Solid Tumors (mRECIST).
7. Performance status (PS) ECOG score ≤1.
8. Child-Pugh score ≤7.
9. Subjects voluntarily participate in this study, and sign the informed consent form, cooperate with the follow-up
10. Adequate organ function, defined as: Hb ≥ 90 g/dL; Neu ≥ 1.5 x 10 ^ 9/L; PLT ≥ 75 x 10 ^ 9/L; ALB ≥2.8 g/dL; TBIL ≤2 times the upper limit of normal; AST and ALT ≤ 3 times the upper limit of normal; Cre ≤1.5 x upper limit of normal; APTT≤1.5 times the upper limit of normal.

Exclusion Criteria:

1. Pathologically confirmed diagnosis of fibrolamellar HCC, sarcomatoid HCC, hepatocellular carcinoma-intrahepatic cholangiocarcinoma (HCC-ICC) mixed type;
2. Previous liver transplantation;
3. History of other malignancies;
4. Previous history of severe mental illness;
5. Uncontrollable hepatic encephalopathy, hepatorenal syndrome, ascites, pleural effusion or pericardial effusion;
6. Active bleeding or coagulation abnormalities, bleeding tendency or receiving thrombolytic, anticoagulant or antiplatelet therapy;
7. Other reasons were judged by the investigator to be unable to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | After the first HAIC treatment, until the disease progresses or dies (during the treatment of the patient) or the toxicity is intolerable，through study completion, an average of 12 months
  The proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including cases of complete remission (CR), partial remission (PR) under mRECIST criteria

SECONDARY OUTCOMES:
Progression-free survival | From date of the first HAIC treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  The date from the date of admission to the date of the first progression of disease or death of any cause.
Overall survival | Through study completion, up to 24 months
  The date from the date of admission to the date of death of any cause
Disease control rate | From date of the first HAIC treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  The percentage of confirmed cases including complete remission (CR), partial remission (PR) and disease stability (SD) among patients with evaluable efficacy
Adverse Events | Until the last medication for 30 days (±7 days) or before the start of other anti-tumor therapy (whichever occurs first).
  Categorized according to NCI Common Toxicity Criteria version 5.0. Summarized in terms of type, severity (grade 1-5), and dose level in tabular format.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Chen, Principal Investigator — 106 Second Zhongshan Road, Guangzhou, Guangdong
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China